CLINICAL TRIAL: NCT05846737
Title: Safety and Efficiency of BCMA CAR-T Cell Therapy in High-risk NDMM Patients With Positive MRD After First-line ASCT: a Prospective, Single-arm, Single-center, Phase II Study.
Brief Title: BCMA CAR-T Cell Therapy in High-risk NDMM Patients With Positive MRD After First-line ASCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023012
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- BCMA CAR-T in high-risk MM with detectable MRD after first-line ASCT (Experimental): Autologous BCMA-directed CAR-T cells, infusion intravenously at a target dose of 2-4 x 10^6 anti-BCMA CAR+T cells/kg.
  Interventions: Biological: anti-BCMA CAR-T

INTERVENTIONS:
Biological: anti-BCMA CAR-T — Autologous BCMA-directed CAR-T cells, infusion intravenously at a target dose of 2-4 x 10^6 anti-BCMA CAR+T cells/kg.

SUMMARY:
This study is a open-label, single-center Phase 2 study to evaluate the efficacy and safety of BCMA CAR-T Cell Therapy in High-risk NDMM Patients With Positive MRD After First-line ASCT. A total of 40 subjects will be enrolled into this study.

DETAILED DESCRIPTION:
The study is a prospective, single-arm, single-centre, phase II study designed to evaluate the efficacy and safety of BCMA CAR-T Cell Therapy in High-risk NDMM Patients With Positive MRD After First-line ASCT. Patients with detectable MRD after undergoing ASCT MRD will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Participants with documented NDMM according to IMWG diagnostic criteria.
3. High-risk MM, as determined by R2-ISS（J Clin Oncol, 2022,40(29):3406-3418.）, Stage III or Stage IV.
4. Has received 3 to 6 cycles of induction therapy, followed by conditioning regimen and ASCT.
5. Screening must be completed within 100 days of ASCT.
6. For subjects receiving consolidation therapy after ASCT, screening must be completed within 60 days after consolidation therapy, and within 6 months after ASCT.
7. Detectable MRD using EuroFlow or NGS, at 100 days after ASCT (minimum sensitivity of 10-5).
8. All screening blood biochemistry: tests should be performed according to the protocol and within 14 days before enrollment. Screening laboratory values must meet the following criteria: a.TBIL<1.5 x upper limit of normal (ULN) (<3 x ULN in patients with Gilbert's syndrome); b.AST and ALT <3 x ULN.; c. Creatinine clearance > 60mL/min (calculated using the Cockroft-Gault formula).
9. Routine blood tests (performed within 7 days, no RBC transfusion, no G-CSF/GM-CSF/platelet agonists, no drug correction within 14 days before screening, no PLT transfusion within 7 days) : WBC ≥ 1.5 x 109/L, ANC ≥ 1.0 x 109/L, Hb ≥ 85 g/L PLT ≥ 75 x 109/L (if BMPC < 50%) or PLT ≥ 50 x 109/L (if BMPC ≥ 50%).
10. Patients must be able to take prophylactic anticoagulant therapy as recommended by the study.
11. The woman is not breastfeeding, is not pregnant and agrees not to be pregnant during the study period and for the following 12 months. Male patients agreed that their spouse would not become pregnant during the study period and for 12 months thereafter.

Exclusion Criteria:

1. Primary plasma cell leukemia.
2. Documented active amyloidosis.
3. Multiple myeloma with central nervous system (CNS) invasion.
4. Has received maintenance therapy.
5. Prior exposure to any BCMA-targeted therapy or CAR-T therapy.
6. Patients with peripheral neuropathy greater than grade 2 or peripheral neuropathy greater than grade 2 with pain at baseline, regardless of whether they were currently receiving medical therapy.
7. Known intolerance, hypersensitivity, or contraindication to BCMA-CART cellular products.
8. Seropositive for human immunodeficiency virus (HIV).
9. Hepatitis B infection.
10. Hepatitis C infection.
11. Life expectancy of <3 months.
12. Women who are pregnant or breastfeeding.
13. Subjects had major surgery within 2 weeks before randomization (for example, general anesthesia), or is not fully recovered from the surgery, or surgery is arranged during study period.
14. Received live attenuated vaccine within 4 weeks prior to study treatment.
15. According to the researcher's judgment, any condition including but not limited to serious mental illness, medical illness, or other symptoms/conditions that may affect study treatment, compliance, or the capability of providing informed consent.
16. Necessary medication or supportive therapy is contraindicated with study treatment.
17. Any diseases or complications that may interfere with the study.
18. Patients are not willing to or cannot comply with study scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Up to 2 year
  The incidence of treatment-emergent adverse events (TEAEs)
MRD-negativity rate | 3 months after CAR-T cell infusion
  Achieving undetectable MRD, as determined by NGF/NGS 3 months after CAR-T cell infusion

SECONDARY OUTCOMES:
Complete response rate (CRR) | 1 month after the CAR-T cell transfusion, after consolidation therapy
  CR or better is defined as percentage of participants who achieve a CR response or Stringent Complete Response (sCR) response accoording to the IMWG criteria
Progression free survival (PFS) | Up to 2 year
  Progression free survival is defined as the time from the date of diagnosis to the date of first documented PD, as defined in the IMWG criteria, or death due to any cause, whichever occurs first
Overall Survival (OS) | Up to 5 year
  Overall survival is measured from the date of diagnosis to the date of the participant's death.

OTHER OUTCOMES:
The CART cell duration in vivo | Up to 1 year
  The copies of BCMA-CART DNA in peripheral blood with qPCR method

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No